CLINICAL TRIAL: NCT01287429
Title: Lung Ultrasound for Acute Dyspnea in Emergency Department - Prospective Multicenter Study on Accuracy, Reproducibility, and Diagnostic Impact of Lung Ultrasound in the Evaluation of Patients With Dyspnea in the Emergency Department
Brief Title: Lung Ultrasound for Acute Dyspnea in Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: Azienda Ospedaliera San Giovanni Battista (Other); San Luigi Gonzaga Hospital (Other); Agnelli Hospital, Italy (Other); Azienda Ospedaliera Ordine Mauriziano di Torino (Other); Martini Hospital, Turin, Italy (Other); Ospedale Cardinal Massaia (Other); Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Emanuele Pivetta, Cancer Epidemiology Unit - University of Turin
Other Study IDs: CEU-UTurin-001
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2010-10

CONDITIONS: Dyspnea; Congestive Heart Failure
Keywords: Ultrasonography
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute dyspnea
  Interventions: Other: lung and pleural ultrasound

INTERVENTIONS:
Other: lung and pleural ultrasound — After the initial diagnostic work-out (medical history, physical examination, EKG, arterious blood gas), the emergency physician will classify dyspnoea in cardiogenic or respiratory dyspnoea and write it down in a specific form (clinical form). Immediately after this, lung and pleural ultrasound will be performed: the physician will describe it and evaluate the etiology again (integrated evaluation form). Then a chest X-ray evaluation will be performed for each patient.

SUMMARY:
Dyspnea is a frequent symptom in patients admitted to the Emergency Department (ED); discriminating between cardiogenic and non-cardiogenic dyspnea is a common clinical dilemma. The initial diagnostic work-out is often not very accurate in defining the etiology and the underlying pathophysiology. In the last years, lung ultrasound (US) has emerged as a useful real-time bedside diagnostic tool in the critical patient. The aim of this study was to evaluate the accuracy, reproducibility, and diagnostic impact of pleural and lung US, performed by emergency physicians at the time of patient first presentation to the ED, in identifying cardiac causes of acute dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to present to the ED with a principal complaint of shortness of breath, deﬁned as either the sudden onset of dyspnea with no history of chronic dyspnea or an increase in the severity of chronic dyspnea in the last 48 hours;
* Presence of an emergency physician with lung US experience at the time of enrollment;
* US examination within 30 minutes after the start of the clinical evaluation.

Exclusion Criteria:

* Dyspnea cases clearly due to neither cardiogenic nor respiratory etiology will considered not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Emergency Departments sample
Sampling Method: Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Pivetta, Principal Investigator — Cancer Epidemiology Unit - University of Turin
Locations (7):
- Italy (7):
  - Emergency Department - AOU San Giovanni Battista, Turin, Italy
  - Emergency Medicine & Surgery Unit - Cardinal Massaia Hospital, Asti
  - Emergency Department - AO Santa Croce e Carle, Cuneo
  - Emergency Medicine Unit - AOU San Luigi Gonzaga, Orbassano
  - Emergency Medicine & Surgery Unit - Pinerolo General Hospital, ASL TO 3, Pinerolo
  - Emergency Medicine and Surgery Unit- AO Mauriziano, Turin
  - Emergency Medicine & Surgery Unit - Martini Hospital, ASL TO 2, Turin

REFERENCES:
- [Background] Ray P, Birolleau S, Lefort Y, Becquemin MH, Beigelman C, Isnard R, Teixeira A, Arthaud M, Riou B, Boddaert J. Acute respiratory failure in the elderly: etiology, emergency diagnosis and prognosis. Crit Care. 2006;10(3):R82. doi: 10.1186/cc4926. Epub 2006 May 24. PMID 16723034
- [Background] Dao Q, Krishnaswamy P, Kazanegra R, Harrison A, Amirnovin R, Lenert L, Clopton P, Alberto J, Hlavin P, Maisel AS. Utility of B-type natriuretic peptide in the diagnosis of congestive heart failure in an urgent-care setting. J Am Coll Cardiol. 2001 Feb;37(2):379-85. doi: 10.1016/s0735-1097(00)01156-6. PMID 11216950
- [Background] Siefkin AD. Dyspnea in the elderly: cardiac or pulmonary? Geriatrics. 1985 May;40(5):63-5, 68-70, 73. PMID 3988043
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404
- [Background] Incalzi RA, Fuso L, Serra M, Basso S, Carosella L, Tramaglino LM, Pistelli R, Carbonin P. Exacerbated chronic obstructive pulmonary disease: a frequently unrecognized condition. J Intern Med. 2002 Jul;252(1):48-55. doi: 10.1046/j.1365-2796.2002.01005.x. PMID 12074738
- [Background] Wang CS, FitzGerald JM, Schulzer M, Mak E, Ayas NT. Does this dyspneic patient in the emergency department have congestive heart failure? JAMA. 2005 Oct 19;294(15):1944-56. doi: 10.1001/jama.294.15.1944. PMID 16234501
- [Background] Fagan TJ. Letter: Nomogram for Bayes's theorem. N Engl J Med. 1975 Jul 31;293(5):257. doi: 10.1056/NEJM197507312930513. No abstract available. PMID 1143310
- [Background] Sackett DL, Straus S. On some clinically useful measures of the accuracy of diagnostic tests. ACP J Club. 1998 Sep-Oct;129(2):A17-9. No abstract available. PMID 9749135
- [Background] Collins SP, Lindsell CJ, Storrow AB, Abraham WT; ADHERE Scientific Advisory Committee, Investigators and Study Group. Prevalence of negative chest radiography results in the emergency department patient with decompensated heart failure. Ann Emerg Med. 2006 Jan;47(1):13-8. doi: 10.1016/j.annemergmed.2005.04.003. Epub 2005 Jun 20. PMID 16387212
- [Background] Kataoka H, Takada S. The role of thoracic ultrasonography for evaluation of patients with decompensated chronic heart failure. J Am Coll Cardiol. 2000 May;35(6):1638-46. doi: 10.1016/s0735-1097(00)00602-1. PMID 10807471
- [Background] Lichtenstein D, Meziere G. A lung ultrasound sign allowing bedside distinction between pulmonary edema and COPD: the comet-tail artifact. Intensive Care Med. 1998 Dec;24(12):1331-4. doi: 10.1007/s001340050771. PMID 9885889
- [Background] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Background] Cardinale L, Volpicelli G, Binello F, Garofalo G, Priola SM, Veltri A, Fava C. Clinical application of lung ultrasound in patients with acute dyspnea: differential diagnosis between cardiogenic and pulmonary causes. Radiol Med. 2009 Oct;114(7):1053-64. doi: 10.1007/s11547-009-0451-1. Epub 2009 Aug 20. PMID 19697100
- [Background] Copetti R, Soldati G, Copetti P. Chest sonography: a useful tool to differentiate acute cardiogenic pulmonary edema from acute respiratory distress syndrome. Cardiovasc Ultrasound. 2008 Apr 29;6:16. doi: 10.1186/1476-7120-6-16. PMID 18442425
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Lichtenstein DA. Ultrasound in the management of thoracic disease. Crit Care Med. 2007 May;35(5 Suppl):S250-61. doi: 10.1097/01.CCM.0000260674.60761.85. PMID 17446785
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Picano E, Frassi F, Agricola E, Gligorova S, Gargani L, Mottola G. Ultrasound lung comets: a clinically useful sign of extravascular lung water. J Am Soc Echocardiogr. 2006 Mar;19(3):356-63. doi: 10.1016/j.echo.2005.05.019. PMID 16500505
- [Background] Reissig A, Kroegel C. Transthoracic sonography of diffuse parenchymal lung disease: the role of comet tail artifacts. J Ultrasound Med. 2003 Feb;22(2):173-80. doi: 10.7863/jum.2003.22.2.173. PMID 12562122
- [Background] Volpicelli G, Cardinale L, Garofalo G, Veltri A. Usefulness of lung ultrasound in the bedside distinction between pulmonary edema and exacerbation of COPD. Emerg Radiol. 2008 May;15(3):145-51. doi: 10.1007/s10140-008-0701-x. Epub 2008 Jan 31. PMID 18236088
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Background] Liteplo AS, Marill KA, Villen T, Miller RM, Murray AF, Croft PE, Capp R, Noble VE. Emergency thoracic ultrasound in the differentiation of the etiology of shortness of breath (ETUDES): sonographic B-lines and N-terminal pro-brain-type natriuretic peptide in diagnosing congestive heart failure. Acad Emerg Med. 2009 Mar;16(3):201-10. doi: 10.1111/j.1553-2712.2008.00347.x. Epub 2009 Jan 29. PMID 19183402
- [Derived] Pivetta E, Goffi A, Lupia E, Tizzani M, Porrino G, Ferreri E, Volpicelli G, Balzaretti P, Banderali A, Iacobucci A, Locatelli S, Casoli G, Stone MB, Maule MM, Baldi I, Merletti F, Cibinel GA, Baron P, Battista S, Buonafede G, Busso V, Conterno A, Del Rizzo P, Ferrera P, Pecetto PF, Moiraghi C, Morello F, Steri F, Ciccone G, Calasso C, Caserta MA, Civita M, Condo' C, D'Alessandro V, Del Colle S, Ferrero S, Griot G, Laurita E, Lazzero A, Lo Curto F, Michelazzo M, Nicosia V, Palmari N, Ricchiardi A, Rolfo A, Rostagno R, Bar F, Boero E, Frascisco M, Micossi I, Mussa A, Stefanone V, Agricola R, Cordero G, Corradi F, Runzo C, Soragna A, Sciullo D, Vercillo D, Allione A, Artana N, Corsini F, Dutto L, Lauria G, Morgillo T, Tartaglino B, Bergandi D, Cassetta I, Masera C, Garrone M, Ghiselli G, Ausiello L, Barutta L, Bernardi E, Bono A, Forno D, Lamorte A, Lison D, Lorenzati B, Maggio E, Masi I, Maggiorotto M, Novelli G, Panero F, Perotto M, Ravazzoli M, Saglio E, Soardo F, Tizzani A, Tizzani P, Tullio M, Ulla M, Romagnoli E; SIMEU Group for Lung Ultrasound in the Emergency Department in Piedmont. Lung Ultrasound-Implemented Diagnosis of Acute Decompensated Heart Failure in the ED: A SIMEU Multicenter Study. Chest. 2015 Jul;148(1):202-210. doi: 10.1378/chest.14-2608. PMID 25654562